CLINICAL TRIAL: NCT01693003
Title: Randomized, Open-label, Crossover Clinical Trial to Assess the Effects of Indacaterol 150 µg d.o. Compared to Tiotropium Bromide 5 µg d.o. on Dyspnea, Dynamic Pulmonary Hyperinflation and Exercise Tolerance in Patients With Moderate COPD
Brief Title: Indacaterol Versus Tiotropium on Dynamic Hyperinflation in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Paulo J Z Teixeira, Clinical professor and chair of the study, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISCMPALABAtrial
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol first (Experimental): Indacaterol 150 µg d.o. during the first 3-week period followed by other 3-week period of tiotropium bromide 5 µg d.o. separated by a "wash-out" phase of at least 5 to 14 days between each treatment period
  Interventions: Drug: Indacaterol; Drug: Tiotropium
- Tiotropium first (Experimental): Tiotropium bromide 5 µg d.o. during the first 3-week period followed by other 3-week period of Indacaterol 150 µg d.o. separated by a "wash-out" phase of at least 5 to 14 days between each treatment period
  Interventions: Drug: Indacaterol; Drug: Tiotropium

INTERVENTIONS:
Drug: Indacaterol — 150 µg d.o. during the first 3 weeks
  Other Names: Onbrez Breezhaler®
Drug: Tiotropium — 150 µg d.o. during 3 weeks
  Other Names: Spiriva Respimat®

SUMMARY:
Exercise intolerance is a major complain of patients with chronic obstructive pulmonary disease (COPD). Dynamic hyperinflation has been recognized as an important limiting factor responsible for the appearance of intolerable dyspnea during exercise. Regular treatment with long-acting bronchodilators promotes a more sustained reduction of hyperinflation and consequent symptom relief and increase in the patient's ability to overcome physical demands of daily life. Tiotropium bromide (TIO) is a new generation, long-acting anticholinergic bronchodilator that significantly improves lung function, reduces symptoms and improves exercise tolerance in patients with advanced COPD. Indacaterol is a new ultra-long duration (>24 h) β2-agonist, which promotes sustained dilation of the bronchi with a once-daily administration. Compared to tiotropium, indacaterol provides evidence that is as effective as tiotropium for bronchodilation, as well as other clinical outcomes such as dyspnea and state of health. However, comparative effects of indacaterol versus tiotropium with regard to outcomes in tolerance, dyspnea and dynamic lung hyperinflation during exercise is scarce. We hypothesized that indacaterol and TIO are not different in terms of exercise tolerance and its determinants (dynamic hyperinflation and dyspnea).

ELIGIBILITY:
Inclusion Criteria:

* Men and women (neither pregnant nor nursing women) ≥40 years of age, with a history of smoking (>20 years/pack) and COPD diagnosis according to GOLD criteria.
* Post-bronchodilator FEV1 >50% and <80%, and FEV1/FVC ≤70% of predicted value.

Exclusion Criteria:

* Hospital admission due to COPD exacerbation or lung infection in the 6 weeks prior to screening, diagnosis of current or previous bronchial asthma, history of allergic rhinitis or other atopic diseases, or peripheral eosinophilia >400/mm3.
* Inability to discontinue the usual bronchodilator therapy prior to initial screening tests, need for continuous oxygen therapy, or arterial oxygen saturation <85% at rest, or history of adverse reactions to sympathomimetic amines or use of inhaled medication.
* Anemia, hypo- or hyperthyroidism, hyperadrenergic conditions, uncontrolled insulin-dependent diabetes mellitus, malignancy, or any disease or condition that limits exercise capacity other than COPD.
* History of drug or alcohol abuse, poor adherence to drug treatment, or treatment with any investigational drug in the month before screening.
* Patients with ventricular arrhythmia.
* Patients with <80% oxyhemoglobin saturation during exercise testing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 3 weeks
  Time between beginning of high intensity constant load (75-85% of the peak achieved in a previous cycloergometer incremental test) cardiopulmonary exercise test and point at which patient cannot tolerate the effort any longer.

SECONDARY OUTCOMES:
Effort-related dyspnea during daily activities | 3 weeks
Airway diameter and volume, and extension of pulmonary emphysema by multidetector helical chest computed tomography | 3 weeks
Oxidative stress before and after exercise tests | 3 weeks
Exercise dyspnea | 3 weeks
  Dyspnea evaluated by Borg scale each 2 minutes during high intensity constant load cardiopulmonary exercise test until exhaustion (peak exercise)
Dynamic pulmonary hyperinflation | 3 weeks
  Inspiratory capacity measured each 2 minutes during high intensity constant load cardiopulmonary exercise test until exhaustion (peak exercise).

OTHER OUTCOMES:
Adverse events | Participants will register adverse events in clinical research diaries or communicate to investigator during 3-week treatment period
  Adverse events, including serious adverse events, will be collected and reported in the CRF (Clinical Research File) of the study.
  Adverse event is any sign, symptom or undesired medical condition that occurs after the beginning of the study even if said event is not considered related to the drug (or therapy) of study. Information on adverse events either reported voluntarily by the patient, identified through questioning by the investigator, or detected by physical examination, laboratory testing or otherwise, will be collected and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Z Teixeira, MD, Study Chair — Santa Casa de Porto Alegre
Locations (1):
- Pavilhão Pereira Filho, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Berton DC, Santos AH, Bohn I Jr, Lima RQ, Breda V, Teixeira PJ. Effects of indacaterol versus tiotropium on exercise tolerance in patients with moderate COPD: a pilot randomized crossover study. J Bras Pneumol. 2016 Sep-Oct;42(5):367-373. doi: 10.1590/S1806-37562015000000334. PMID 27812637